CLINICAL TRIAL: NCT01499524
Title: A Longitudinal Study of Alterations in Metabolic Markers and Gut Hormones in Pregnant and Non-pregnant Patients With Intrahepatic Cholestasis of Pregnancy, Gestational Diabetes Mellitus and Normal Pregnant and Non-pregnant Controls
Brief Title: The Metabolic Profile in Intrahepatic Cholestasis of Pregnancy and Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: JROHH0280
Record Dates: First submitted 2011-09-26; First posted 2011-12-26 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Intrahepatic Cholestasis of Pregnancy; Gestational Diabetes Mellitus
Keywords: ICP, GDM
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, whole blood, plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ICP is known to cause abnormal bile acid homeostasis and to be associated with an increased risk of diseases of the biliary system in later life. There have been small studies (Dann et al. 2006; Wójcicka-Jagodzińska et al. 1989) suggesting that it causes dyslipidaemia (raised lipids) and impaired glucose tolerance in pregnancy. However the underlying mechanisms of these abnormalities is not known. Similarly the influence of cholestasis on fetal metabolism is not known, and nor is the role of the placenta. It is also not known whether women with ICP have a predisposition to abnormal lipid and glucose homeostasis when they are not pregnant.

GDM is characterized by raised plasma glucose levels in pregnant women (in the absence of pre-pregnancy diabetes mellitus). This condition is associated with large-for-gestational age babies and obstructed labour. Women with GDM have increased risk of subsequent type 2 diabetes mellitus, and if they have this condition in a subsequent pregnancy there is an increased risk of stillbirth. This work is important to understand the causes of the metabolic abnormalities associated with ICP and GDM. If we demonstrate abnormal lipid and glucose profiles, these may be of relevance to the fetal complications of both disorders. It will also be of relevance to the future health of affected women and their children.

DETAILED DESCRIPTION:
CLINICAL FEATURES OF INTRAHEPATIC CHOLESTASIS OF PREGNANCY:

Intrahepatic cholestasis of pregnancy (ICP), is a pregnancy-specific liver disorder which typically presents with maternal pruritus (itching) in late pregnancy and affects about 0.7% of women in the UK. Biochemically, it is characterised by liver dysfunction with raised serum bile acids, and clinically by a significantly increased incidence of fetal complications, including spontaneous preterm labour, fetal distress, meconium staining of the amniotic fluid and sudden fetal death (Geenes and Williamson 2009).

The cause of ICP is complex and not fully understood. In addition the pathological mechanisms behind the adverse fetal outcomes have not been elucidated. The maternal disease is likely to be caused by interaction between sex hormone metabolites and bile acids in genetically susceptible women (Abu-Hayyeh et al. 2010). To date, we and others have identified genetic variation in several biliary transporters e.g. ABCB4, ATP8B1, ABCB11 and the main bile acid receptor, FXR, that predispose women to the disease (Dixon et al., 2000; Mullenbach et al., 2005; Pauli-Magnus et al., 2004; Van Mil et al, 2007; Dixon et al. 2009). Due to their inherent toxicity, bile acids are also likely to be responsible for the fetal component of the disease. Consistent with this the incidence of fetal complications has been shown to be increased in pregnancies where the levels exceed 40 uMol /L (Glantz et al., 2004). There are currently several theories about how bile acids may affect fetal wellbeing; with regard to the increased incidence of spontaneous prematurity, they have been shown to cause premature delivery in sheep (Campos et al., 1986), and increased myometrial contractility in response to oxytocin (Germain et al., 2003; Israel et al., 1986). Furthermore, bile acids are also known to cause increased colonic motility in rabbits (Snape et al., 1980) and cardiac dysrhythmias in rats (Williamson et al., 2001), which could explain meconium staining of the amniotic fluid and sudden fetal death respectively. While it is known that bile acids can be transported by proteins in the placenta, the precise role of the placenta in bile, lipid and glucose metabolism is not known. Our group has demonstrated that cholestasis alters lipid pathways in mouse placentas (unpublished data) but this has not been studied in humans.

BILE ACID HOMEOSTASIS:

Bile acids are the end product of hepatic cholesterol metabolism and act as the main route of excretion for cholesterol. In the adult human two primary bile acids are produced by the liver, i.e. cholic acid and chenodeoxycholic acid. There is some evidence that maternal bile acids gradually rise with advancing gestation, but they usually remain within normal limits (< 14 uMol /L) (Fulton et al., 1983; Pascual et al., 2002). This is in contrast to an ICP pregnancy, where maternal bile acids may be raised to 100 times the upper limit of normal (Walker et al.,2002). In OC, elevated levels of bile acids are also found in the fetal circulation (Laatikainen, 1975).

THE ROLE OF BILE ACIDS IN LIPID AND GLUCOSE METABOLISM:

There is accumulating evidence that FXR, the nuclear hormone receptor responsible for regulation of bile acid homeostasis, also plays a role in the regulation of lipid and glucose metabolism. FXR null mice have been shown to have abnormal blood lipid profiles including elevated plasma cholesterol, low density lipoprotein, high density lipoprotein and triglyceride levels (Ma, 2006). They also exhibit glucose intolerance and reduced insulin sensitivity (Zhang, 2006). Furthermore, ICP patients have raised levels of cholesterol and other lipid parameters (Dann et al. 2006). Specifically, the serum concentrations of low-density lipoprotein (LDL), apolipoprotein B-100, cholesterol and total cholesterol were markedly increased in women with ICP. They have also been shown to have impaired glucose tolerance (Wójcicka-Jagodzińska et al. 1989). Recent data from our group (Martineau et al. 2014, 2015) and others (Marschall et al. 2014) have shown that women with ICP have increased rates of GDM, and implicate raised serum bile acids in susceptibility to diabetes mellitus. Therefore this study will also include women with ICP and superimposed GDM in addition to women with GDM in the absence of ICP. This will enable us to evaluate the impact of cholestasis on the onset of diabetes mellitus in pregnant women.

In cholestasis bile acids accumulate in the liver, and this results in the induction of pathways that enhance bile acid excretion. This may also cause abnormal cholesterol and triglyceride levels. Bile acids also signal via FXR in the gut. Bile acids are stored in the gallbladder in the fasting state and released following ingestion of a meal. Once bile acids are in the intestine they are transported into enterocytes (gut cells) where they activate FXR which causes production and release of the hormone FGF19. FGF19 binds the FGF4 receptor on hepatocytes, and signals (via the jnk kinase pathway) to suppress cholesterol 7 alpha-hydroxylase (CYP7A1), a critical rate-limiting enzyme in synthesis of bile acids from cholesterol. There have been no studies of the gut-liver axis in pregnancy, but we hypothesise that abnormal bile acid signalling causes raised cholesterol in addition to increased serum bile acids.

Bile acids also bind the G-protein-coupled receptor (TGR5). In the gut this results in release of glucagon-like peptide-1 (GLP-1)(Thomas et al. 2009). GLP-1 is an anti-diabetic hormone that increases glucose-dependent insulin production and decreases glucagon production by the pancreas. To date, there have been no studies of the relationship between cholestasis and GDM and the levels of other fasting gut hormones that may influence glucose and lipid metabolism in pregnancy.

ELIGIBILITY:
Inclusion criteria:

* Women with intrahepatic cholestasis of pregnancy, defined as pruritus in pregnancy in association with raised serum bile acids and in the absence of an alternative cause.
* Women with gestational diabetes mellitus (GDM) according to the diagnostic criteria used at the referring centre
* Non-pregnant parous females with previous ICP or GDM.
* Women who are able to give consent.
* Women >16 and <70 years of age. Controls
* Pregnant women not affected by ICP or GDM .
* Non-pregnant parous females with previous uncomplicated pregnancy.
* Women who are able to give consent.
* Women >16 and <70 years of age.

Exclusion Criteria

* Males.
* Non-pregnant females with other medical disorders that can cause liver impairment, abnormal lipid or glucose metabolism in pregnancy, e.g. pre-eclampsia, acute fatty liver of pregnancy, pre-existing diabetes mellitus
* Pregnant females with a history of other medical disorders that can cause liver impairment, abnormal lipid or glucose metabolism in pregnancy, e.g. pre-eclampsia, acute fatty liver of pregnancy, pre-existing diabetes mellitus
* Women who are not able to give consent.
* Women <16 and >70 years of age.

Ages: 16 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women age 16-70
Study Population: Pregnant and non pregnant women who have had intrahepatic cholestasis of pregnancy and/or gestational diabetes mellitus matched with parous women who have had uncomplicated pregnancies
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2011-11; Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
To establish whether raised serum bile acids are associated with abnormalities in cholesterol and triglycerides in the mother and fetus mother and fetus. | 5 years
  Maternal serum samples from women with ICP and controls will be collected to measure cholesterol and triglycerides

SECONDARY OUTCOMES:
To establish the relationship between raised serum bile acids in the mother and fetus and abnormalities in: Glucose homeostasis, gut liver signaling hormones related to FGF 19, glucose and C4 levels, Gut hormone secretion | 5 years
  Maternal serum samples from women with ICP and controls will be collected to measure FGF 19 and glucose

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Williamson, MBChBMDFRCP, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Guy's & St Thomas' NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust Hammersmith, London

IPD SHARING:
Plan to Share IPD: No
Any results and findings will be disseminated in research publications.

REFERENCES:
- [Result] Mitchell AL, Ovadia C, Syngelaki A, Souretis K, Martineau M, Girling J, Vasavan T, Fan HM, Seed PT, Chambers J, Walters J, Nicolaides K, Williamson C. Re-evaluating diagnostic thresholds for intrahepatic cholestasis of pregnancy: case-control and cohort study. BJOG. 2021 Sep;128(10):1635-1644. doi: 10.1111/1471-0528.16669. Epub 2021 Apr 6. PMID 33586324
- See also: Re-evaluating diagnostic thresholds for intrahepatic cholestasis of pregnancy: case-control and cohort study — https://pubmed.ncbi.nlm.nih.gov/33586324/

DOCUMENTS (1):
  • Study Protocol (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT01499524/Prot_000.pdf